CLINICAL TRIAL: NCT06626282
Title: PReserving Fertility and Quality of Life IN Belgian Female Paediatric CancEr SurvivorS
Brief Title: Fertility and Ovarian Reserve in Female Childhood Cancer Survivors
Acronym: PRINCESS
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Liege (Other)
Collaborators: La Fondation contre le cancer, Belgique (Unknown)
Responsible Party: Principal Investigator, Bianca David, MD, Centre Hospitalier Universitaire de Liege
Other Study IDs: OST 2022/2173; 2023/388 (Other: Central Ethical Committee from CHULiege); B7072023000101 (Other: Belgian EudraCT Number)
Record Dates: First submitted 2024-10-02; First posted 2024-10-03 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Childhood Cancer Survivors; Fertility; Ovarian Reserve; CED; Ovarian Reserve Markers; Cryopreservation; Alkylating Agents; Female

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples With DNA — EDTA tubes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Ovarian function impairment affects the quality of life of the survivors of paediatric cancer by impacting fertility, bone quality and mental and cognitive health. The objective of this project is to evaluate the impact of low-intermediate dose alkylating agents associated or not with ovarian cryopreservation technique on ovarian function in female survivors of paediatric cancer. We propose to identify new epigenetic markers in order to predict the risk of premature ovarian insufficiency. The project will be led by a national multi-disciplinary team (paediatric oncologists, gynaecologists, endocrinologists). Paediatric cancer clinical data (therapy, fertility preservation, ...) will be extracted from the Paediatrics Late Effects database and additional data will be collected during PRINCESS fertility evaluation. Through translational and multi-disciplinary approaches, results should improve quality of life and fertility preservation in female survivors of paediatric cancer by developing new personalised screening tools for premature ovarian insufficiency.

DETAILED DESCRIPTION:
A. Objectives:

In a cohort of female survivors of paediatric cancer aged of at least 18 years old at the time of evaluation, the main objectives of the project PRINCESS are:

1. to evaluate the impact of low-intermediate dose alkylating agents on ovarian function and fertility;
2. to assess the impact of ovarian tissue cryopreservation, used as fertility preservation technique, on further ovarian function and fertility;
3. to identify new screening tools of premature ovarian insufficiency, using targeted and whole genome methylation techniques.

B. Project Design:

The complementarity of the promoters 'and co-applicants skills allows the building of a national translational team which relies on the pre-clinical, clinical and research expertise of paediatric oncologists (Drs Dedeken, De Ville de Goyet and Piette), endocrinologist (Dre Parent) and gynaecologists (Drs Demeestere, Dolmans, Henry and Jadoul). The promoter and co-promotor will directly supervise Dr Bianca David (PhD student) who will contribute to all aspects of the research. The PhD student will be hosted in the LBTD/GIGA-Cancer/Neurosciences and will benefit from its infrastructure, the help of technicians and the expertise of the AS Parent team for epigenetic studies.

Participants eligible to participate to the PRINCESS project (n=170) and controls (n=170) will be invited by a coordinating nurse to take part to PRINCESS fertility evaluation in the medically assisted reproduction centre of one of the three participating institutions. During the first consultation, the PRINCESS project will be explained to the participants, who will sign an informed consent. The expert, with the help of the coordinating nurse, will present the PRINCESS questionnaire including information about their fertility and parenthood situation to the participant, who will then complete it in privacy. A second consultation will take place after minimum 6 weeks without hormonal contraception and ideally between day 2-5 of the menstrual cycle. During this consultation, clinical, biological and ultrasound evaluations will be performed (see below, data collection). A third consultation will be organized to inform he participants of their results. Participants will be offered a compensation for participating to the study.

C. Data collection

1. Data extracted from the Paediatrics Late Effects project at first paediatric cancer and/or relapse(s) and/or progression(s) and/or second cancer(s)

   * Type of cancer
   * Dates of diagnosis and end of treatment
   * Treatment details (type and doses of chemotherapy, type and field of radiotherapy, type of surgery, stem cell transplantation)
   * Fertility preservation measures
   * Relevant late effects (endocrine, gynaecology, etc.), defined following the Common Terminology Criteria for Adverse Events, version 4.03 (2010-06-14).
   * Vital status at last news
2. Data collected during PRINCESS fertility evaluation

   * Height, weight, body mass index
   * Puberty history, date of menarche and menstrual cycles history
   * Pregnancies, childbirth, use of hormonal therapies, including contraception,
   * Menopause substitutive hormonal treatment
   * Measurement of LH, FSH, oestradiol, progesterone, prolactin, TSH, T4, AMH levels
   * Evaluation of the ovarian reserve by ultra-sound (antral follicle count).

Note: one blood EDTA tube will be collected from each patient and stored in a bio-bank in CHU of Liege for later epigenetics analysis.

Data collected by PRINCESS questionnaire Marital status Lifestyle (tobacco/cannabis/alcohol consumption) Level of education Occupation For children and adolescent female cancer survivors who ever tried to become pregnant: use of medical help (and type), pregnancy course (live birth with or without birth defect, miscarriage, medical abortion, stillbirth)

ELIGIBILITY:
Inclusion Criteria:

* Child and adolescent female patients included in the Paediatrics Late Effects Project:
* diagnosed with cancer1 between 01/01/2004 and 31/12/2018
* <17 years old at diagnosis
* treated at CHU Liège site Citadelle or CHC, Cliniques Universitaires Saint-Luc and HUDERF
* alive
* ≥ 18 years-old at time of recruitment.

Exclusion Criteria:

* Cancer diagnosis for controls

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — females without hormonal treatment in order to change gender
Study Population: Child and adolescent female patients included in the Paediatrics Late Effects Project.
  Controls will be age-, sex- and socio-economic-matched individuals starting with the siblings of the survivors. Belgian (http://statbel.fgov.be/en) public demographic, socioeconomic and birth registries will be used to exclude any bias in controls recruitment.
Sampling Method: Probability Sample
Enrollment: 340 (Estimated)
Dates: Start 2024-10-09 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
The index of fertility | 2027
  having children among survivors in compared with controls
The rate of menopause and POI | 2027
  Number of participants in POI
The rate of premature or delayed puberty | 2027
  Number of participants with premature/delayed puberty
The rate of negative pregnancy outcome (miscarriage, medical abortion, stillbirth or birth | 2028
  Number of participants with pregnancy problems
The rate of use of medical help to become pregnant among survivors | 2028
  Number of participants using FIV
The rate of irregular menstruation, ovulatory disorders | 2027
  Number of participants with cycle disruptions

CONTACTS AND LOCATIONS:
Locations (3):
- Belgium (3):
  - Hopital de la Citadelle, Liège, Wallonia
  - Cliniques Universitaires Saint-Luc, Brussels
  - HUDERF, Brussels

IPD SHARING:
Plan to Share IPD: No